CLINICAL TRIAL: NCT05827315
Title: Incidence, Impact and Mechanisms of Perioperative Right VEntricular Dysfunction (IMPRoVE)
Acronym: IMPRoVE
Status: Not yet recruiting | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other); Royal London Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Ben Shelley, Honorary Professor/Consultant in Cardiothoracic Anaesthesia and Intensive Care, University of Glasgow
Other Study IDs: 22/ANAES/06
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Right Ventricular Dysfunction
Keywords: Echocardiography; T1 CMR; Major non-cardiac surgery; Perioperative Complication; Postoperative myocardial injury; Right heart catheterisation; Coronary sinus sampling
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Thoracic surgery cohort: 35 patients undergoing thoracic surgery with lung resection and one lung ventilation under primarily general anaesthesia.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: T1 Cardiovascular Magnetic Resonance; Diagnostic Test: Right heart catheterisation and coronary sinus blood sampling
- Upper gastrointestinal surgery cohort: 35 patients undergoing upper gastrointestinal surgery with one lung ventilation under primarily general anaesthesia.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: T1 Cardiovascular Magnetic Resonance
- Colorectal surgery cohort: 35 patients undergoing elective colorectal surgery under primarily general anaesthesia.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: T1 Cardiovascular Magnetic Resonance
- Vascular surgery cohort: 35 patients undergoing elective open abdominal aortic surgery under primarily general anaesthesia.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: T1 Cardiovascular Magnetic Resonance
- Orthopaedic surgery cohort: 35 patients undergoing elective primary hip or knee arthroplasty under spinal anaesthesia +/- sedation.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: T1 Cardiovascular Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography will be performed by BSE accredited echocardiographers in all 175 patients preoperatively and on day 2-4 postoperatively.
Diagnostic Test: T1 Cardiovascular Magnetic Resonance — T1 CMR will be performed in 10 patients from each of the 5 surgical groups (50 patients in total) preoperatively and on day 2-4 postoperatively.
Diagnostic Test: Right heart catheterisation and coronary sinus blood sampling — 10 patients from the thoracic surgical group will undergo right heart catheterisation and coronary sinus blood sampling.
  Groups: Thoracic surgery cohort

SUMMARY:
A study to see how common right heart failure (right ventricular dysfunction) after major surgery is, and to investigate if right ventricular dysfunction causes worse patient outcomes after surgery.

DETAILED DESCRIPTION:
Heart attacks are relatively rare around the time of surgery, however by measuring blood markers of heart injury, recent research has revealed that heart injury which otherwise may not be immediately obvious is common. Whilst this type of heart injury appears to be strongly linked to patient outcomes (complications, recovery and survival), the causes and potential treatments for it are not well understood.

Our research group has specialist knowledge about the right-hand side of the heart (right-heart) - the side that pumps blood through the lungs - which is less commonly considered or studied around the time of surgery. We have shown in previous studies using magnetic resonance imaging (MRI) scans (specialised whole-body scans which use a magnet rather than X-rays), evidence of right-heart function deteriorating after surgery. We want to test the idea that some of the blood marker evidence of heart injury reflects injury to the right-heart and more importantly that we can protect the right-heart around the time of surgery, reducing injury and improving patient outcomes.

We will examine these questions in the following ways:

1. With patients' permission, we will perform detailed ultrasound scans of the heart (echocardiography), and blood measurement of injury markers in 175 patients undergoing different types of major surgery. This will allow us to assess how common heart injury is (visible on scans of both sides of the heart), whether it makes any difference to a patient's outcome and whether it explains the changes seen in blood markers.
2. We will ask 50 of these patients to undergo MRI scans of the heart pre- and post-operatively to allow us to identify evidence of injury resulting from heart inflammation around the time of surgery. Inflammation is common following surgery and occurs throughout a patient's body - we believe heart inflammation may be responsible for postoperative heart injury.
3. In 10 of these patients, we will seek to obtain blood samples from vessels flowing into the heart (easily obtained from a simple blood sample) and from veins flowing out of the heart, obtained by passing a fine tube into the heart via blood vessels in a patient's neck under X-ray guidance. This will allow us to examine what happens to immune cells as they pass through the heart (i.e., are they activated by heart inflammation?) and better understand the meaning of the changes seen on MRI scans.

This study will give us a better understanding of which patients are likely to suffer heart injury around the time of surgery and how this injury occurs. With this knowledge, future patients could receive personalised treatment plans aimed at preventing injury and improving outcomes. We are not testing any new treatments in this study.

ELIGIBILITY:
Main echocardiography study

Inclusion Criteria:

1. Provision of informed consent
2. Age >18 years
3. Planned elective primary hip or knee joint replacement under spinal anaesthesia, major colorectal, major vascular surgery or surgery requiring one lung ventilation with or without lung resection

Exclusion Criteria:

1. Pregnancy
2. On-going participation in any investigational research which could undermine the scientific basis of the study
3. Previous major surgery within three months prior to recruitment
4. Previous participation in the IMPRoVE study at any time
5. Inadequate comprehension of English resulting in inability to comply with instructions while undergoing investigations required for main study and sub-studies.

Additional exclusion criteria applicable to the T1 CMR sub-study includes:

1. Atrial fibrillation at baseline
2. Contraindication to cardiac magnetic resonance imaging (metal work in body etc)
3. Contraindication to IV Gadolinium: acute or chronic renal failure, allergy to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 175 patients of 18 years or older undergoing major non-cardiac surgery in the West of Scotland. Patients will be recruited from the Golden Jubilee National Hospital, Queen Elizabeth University Hospital, and Glasgow Royal Infirmary.
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative Right ventricular dysfunction (RVD) | Echocardiography performed preoperatively and at day 2-4 postoperatively to measure change in RV function
  RVD diagnosed by transthoracic echocardiography, defined as:
  * 2D-speckle tracking derived RV free wall peak longitudinal strain (FWLS) less negative than -20%.
  * Or, (where not available) two of Tricuspid Annular Plane Systolic Excursion (TAPSE) <16mm, S' Wave velocity at the tricuspid annulus <10cm/s or tissue doppler RV index of myocardial performance >0.55
Days alive and at home at 30 days postoperatively (DAH30) | Day 30 postoperatively
  DAH30 is a continuous number between 0 and 30 which reflects, out of the 30 days following surgery, the total number of those days that a patient spends alive and at home. If a patient dies within those 30 days, their value is set to 0. Data for DAH30 will be obtained by follow-up phone calls following the 30th postoperative day.

SECONDARY OUTCOMES:
Incidence of postoperative left ventricular dysfunction (LVD) | Echocardiography performed preoperatively and at day 2-4 postoperatively to measure change in LV function
  LVD classified as mild, moderately or severely impaired, defined by 2D-echocardiography derived biplane LV ejection fraction and the presence of wall motion abnormalities.
Cardiac biomarkers | BNP and troponin measured preoperatively, on postoperative days 1 and 2 and on day of postoperative echocardiography (occurring on postoperative days 2-4).
  Natriuretic peptides and high sensitivity troponin will be measured pre- and postoperatively.
Cardiovascular complications | Day of postoperative echocardiography (day 2-4 postoperatively) and at discharge (on average one week).
  Incidence of myocardial infarction, cardiac death, non-fatal cardiac arrest, coronary revascularisation, pulmonary embolus, deep-veined thrombosis, or new onset atrial fibrillation, and major adverse cardiac events
Renal outcomes | Day of postoperative echocardiography (day 2-4 postoperatively) and at discharge (on average one week).
  Kidney Disease Improving Global Outcome (KDIGO) classification of Acute Kidney Injury (AKI).
Pulmonary outcomes | Day of postoperative echocardiography (day 2-4 postoperatively) and at discharge (on average one week).
  Atelectasis, pneumonia, acute respiratory distress syndrome or pulmonary aspiration
Infection Outcomes | Day of postoperative echocardiography (day 2-4 postoperatively) and at discharge (on average one week).
  Fever and clinical suspicion of infection
Neurological outcomes | Day of postoperative echocardiography (day 2-4 postoperatively) and at discharge (on average one week).
  Delirium and stroke
Sequential Organ Failure Assessment (SOFA) Score | Postoperative day 1,2, day of postoperative echocardiography in all patients. In patients admitted to HDU/ICU, SOFA score will be collected from postoperative day 0-7.
  Score 0-24, where higher scores are a worse outcome.
Fifteen-point Quality of Recovery Score (QoR-15) | Pre-operatively and day of postoperative echocardiography (day 2-4 postoperatively).
  Fifteen questions assessing the quality of a patients recovery, each question is scored 0-10 with higher scores indicating a worse outcome.
World Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0) | Preoperatively, and at day 30, day 90, and one year postoperatively.
  WHODAS 2.0 is a self administered questionnaire that assesses a patient's health and disability. Twelve questions are scored 0-4, where a higher score indicates a worse outcome.
EuroQoL Dimension Health Related Quality of Life Questionnaire (EQ-5D-5L) | Preoperatively, and at day 30, day 90, and one year postoperatively.
  EQ-5D-5L is a self administered questionnaire that assesses 5 dimensions of a patient's quality of life. Each dimension is scored 1-5, where a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Shelley, Principal Investigator — National Waiting Times Centre Board
Locations (3):
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keast T, McErlane J, Kearns R, McKinlay S, Raju I, Watson M, Robertson KE, Berry C, Greenlaw N, Ackland G, McCall P, Shelley B. Study protocol for IMPRoVE: a multicentre prospective observational cohort study of the incidence, impact and mechanisms of perioperative right ventricular dysfunction in non-cardiac surgery. BMJ Open. 2023 Sep 6;13(9):e074687. doi: 10.1136/bmjopen-2023-074687. PMID 37673452